CLINICAL TRIAL: NCT02128958
Title: A Phase 2 Study in the Second-Line Treatment of Advanced Hepatocellular Carcinoma in Subjects With Child-Pugh Class B Cirrhosis
Brief Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled of the Efficacy and Safety of CF102 in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF102-201HCC
Record Dates: First submitted 2014-04-27; First posted 2014-05-01 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Child-Pugh Class B Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CF102 (Experimental): orally q12h
  Interventions: Drug: CF102
- Placebo tablets of CF102 (Placebo Comparator): orally q12h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF102 — orally q12h
  Other Names: IB-MECA
  Arms: CF102
Drug: Placebo — orally q12 hours
  Other Names: Inactive pill
  Arms: Placebo tablets of CF102

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial in subjects with advanced HCC and CPB cirrhosis whose disease has progressed while taking 1 prior systemic drug therapy for HCC.

DETAILED DESCRIPTION:
The trial will evaluate the efficacy and safety of CF102 as compared to placebo. Subjects will be randomly assigned in a 2:1 ratio to treatment with oral doses of either CF102 25 mg or matching placebo administered twice daily (BID) for consecutive, 28-day cycles. Subjects will be evaluated regularly for safety. Tumor imaging will be performed every 8 weeks. Treatment will continue until the subject experiences unacceptable drug-related intolerability. Subjects will return for a follow-up visit 28 days after completion of the last dose of study drug, and every attempt will be made to obtain survival data on all randomized subjects. Subjects who discontinue will be followed indefinitely for survival status. The trial will continue until 75 deaths have been recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Diagnosis of HCC:

   * For subjects without underlying cirrhosis at the time of diagnosis, diagnosis of HCC documented by cytology and/or histology.
   * For subjects with underlying cirrhosis at the time of diagnosis, diagnosis of HCC established according to the American Association for the Study of Liver Diseases Practice Guideline algorithm (Appendix E).
3. HCC is advanced, ie, treatment-refractory or metastatic, and no standard therapies are expected to be curative.
4. Receipt of 1 previous systemic drug therapy for at least 3 weeks and withdrawal from treatment due either to intolerability or to radiographic disease progression. If treatment was withdrawn due to intolerability manifested as a Grade 3 or 4 event by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE v4.0), less than 3 weeks of continuous prior administration prior to withdrawal is acceptable (see also Exclusion Criterion #3).
5. Prior systemic treatment was discontinued for at least 2 weeks prior to the Baseline Visit.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2 (Appendix B).
7. Cirrhosis classified as Child-Pugh Class B (Appendix C).
8. The following laboratory values must be documented within 3 days prior to the first dose of study drug:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Platelet count ≥ 75 × 109/L
   * Serum creatinine ≤ 2.0 mg/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × the upper limit of normal (ULN)
   * Total bilirubin ≤ 3.0 mg/dL
   * Serum albumin ≥ 2.8 g/dL
   * Prothrombin time (PT) no greater than 6 seconds longer than control.
9. Life expectancy of ≥ 6 weeks.

Exclusion Criteria:

1. Receipt of no, or of >1, prior systemic drug therapies for HCC.
2. Receipt of systemic cancer therapy, immunomodulatory drug therapy, immunosuppressive therapy, or corticosteroids > 20 mg/day prednisone or equivalent within 14 days prior to the Baseline Visit or concurrently during the trial.
3. Presence of an acute or chronic toxicity of prior chemotherapy that has not resolved to ≤ Grade 1, as determined by CTCAE v 4.0.
4. Locoregional treatment within 4 weeks prior to the Baseline Visit.
5. Major surgery or radiation therapy within 4 weeks prior to the Baseline Visit.
6. Use of any investigational agent within 4 weeks prior to the Baseline Visit.
7. Child-Pugh Class A or C cirrhosis, or hepatic encephalopathy.
8. Occurrence of esophageal or other gastrointestinal hemorrhage requiring transfusion within 4 weeks prior to the Baseline Visit.
9. Active bacterial, viral, or fungal infection requiring systemic therapy or operative or radiological intervention.
10. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
11. Liver transplant.
12. Active malignancy other than HCC.
13. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4) (Appendix B).
14. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
15. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females.
16. Pregnant or lactating female.
17. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with trial participation or study drug administration; may interfere with the informed consent process and/or with compliance with the requirements of the trial; or may interfere with the interpretation of trial results and, in the Investigator's opinion, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, Study Director — Can-Fite BioPharma Ltd
Locations (21):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Simmons Cancer Center, Dallas, Texas
- Bulgaria (6):
  - Complex Oncology Center - Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment Central Onco Hospita, Plovdiv
  - Multiprofile Hospital for Active Treatment "Tokuda Hospital Sofia" AD, Sofia
  - Multiprofile Hospital for Active Treatment for women's health - Nadezhda, Sofia
  - Multiprofile Hospital for Active Treatment Serdica, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina" EAD, Varna
- Rabin Medical Center, Petah Tikva, Israel
- Romania (8):
  - Institutul Clinic Fundeni - Sectia Oncologie Medicala, Bucharest
  - Clinica Bendis - Oncologie Medicala, Cluj-Napoca
  - Centrul de Oncologie ONCOLAB, Craiova
  - Institutul Regional de Oncologie Iasi - Sectia Oncologie Medicala, Iași
  - Spitalul Pelican Impex SRL- Sectia Oncologie Medicala, Oradea
  - SC DACMED SRL - Oncologie, Ploieşti
  - Spitalului Clinic Judetean de Urgenta - Sectia Oncologie Medicala, Sibiu
  - Spitalul Judetean de Urgenta "Sf. Ioan Cel Nou" - sectia Oncologie Medicala, Suceava
- Serbia (4):
  - Vojnomedicinska Akademija Beograd, Belgrade
  - Institut za Onkologiju Vojvodine, Kamenitz
  - Zdravstveni Centar Kladovo Služba Onkologije, Kladovo
  - Klinički Centar Niš Klinika za Onkologiju, Niš

REFERENCES:
- [Background] Stemmer SM, Manojlovic NS, Marinca MV, Petrov P, Cherciu N, Ganea D, Ciuleanu TE, Pusca IA, Beg MS, Purcell WT, Croitoru AE, Ilieva RN, Natosevic S, Nita AL, Kalev DN, Harpaz Z, Farbstein M, Silverman MH, Bristol D, Itzhak I, Fishman P. Namodenoson in Advanced Hepatocellular Carcinoma and Child-Pugh B Cirrhosis: Randomized Placebo-Controlled Clinical Trial. Cancers (Basel). 2021 Jan 7;13(2):187. doi: 10.3390/cancers13020187. PMID 33430312

RESULTS

PARTICIPANT FLOW:
Groups:
- CF102: CF102 25 mg capsules administered orally BID
- Placebo Tablets of CF102: Placebo capsules administered orally BID
Period: Overall Study
Arm/Group | CF102 | Placebo Tablets of CF102
Started | 50 | 28
Completed | 29 | 18
Not Completed | 21 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF102 | Placebo Tablets of CF102 | Total
Number analyzed (Participants) | 50 | 28 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.64) | 65.2 (10.22) | 63.4 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 38 | 19 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 48 | 27 | 75
  Black/African | 1 | 0 | 1
  Oriental | 0 | 1 | 1
  Other | 1 | 0 | 1
Diagnostic Procedure [Count of Participants; unit: Participants]
  Cytology/Histology | 27 | 17 | 44
  American Association for the Study of Liver Diseases | 23 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Overall Survival
Description: Evaluate the efficacy of orally administered CF102 25 mg twice daily (BID) as compared to placebo, as determined by Overall Survival (OS), when used as second-line therapy in subjects with advanced hepatocellular carcinoma (HCC) and Child-Pugh Class B (CPB) cirrhosis. Overall Survival is defined as the time from Baseline (Cycle 1 Day 1) to death due to any cause, calculated as (date of death- date of Cycle 1 Day 1) +1.OS will be summarized in months, which will be obtained by dividing OS in days by 30 days/month. Summary statistics will be determined using the Kaplan-Meier (KM) estimate of the survival function and the between-treatment comparison will be performed using the logrank test as the primary analysis.
Time Frame: From date of first treatment (Cycle 1 Day 1) until date of death from any cause, assessed up to 12 months
Population: The analysis of the primary outcome measure was performed on the Intent-To-Treat (ITT) Population, defined as all subjects who received at least one dose of study medication (i.e., Safety Population) with any post-Baseline assessment recorded. Exclusion of subjects from the ITT Population was determined prior to unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
Participants
  12-month Survival - Yes | 16 | 4
  12-month Survival - No | 34 | 24
Statistical Analysis 1: Comparison: CF102 vs Placebo Tablets of CF102; The between-treatment comparison (CF102 vs Placebo) of Overall Survival will be performed using the log rank test as the primary analysis; Test type: Other; p = 0.536, Log Rank

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP) is the time from Baseline to the first Overall Response of Progressive Disease (PD), calculated as date of first PD - date of Cycle 1 Day 1+1. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. TTP will be summarized in months, which will be obtained by dividing TTP in days by 30 days/month. Summary statistics will be determined using the KM estimate of the survival function for TTP. The between-treatment comparison will be performed using the logrank test.
Time Frame: From date of first treatment (Cycle 1 Day 1) until the date of first documented progression, assessed up to 36 months
Population: The analysis of the secondary outcome measure was performed on the Intent-To-Treat (ITT) Population, defined as all subjects who received at least one dose of study medication (i.e., Safety Population) with any post-Baseline assessment recorded. Exclusion of subjects from the ITT Population was determined prior to unblinding.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
Months | 5.1 [1.9 to 11.2] | 3.3 [1.9 to 33.2]
Statistical Analysis 1: Comparison: CF102 vs Placebo Tablets of CF102; The between-treatment comparison (CF102 vs Placebo) of Time to Progression will be performed using the log rank test as the primary analysis; Test type: Other; p = .371, Log Rank

3. Secondary Outcome: Time to Progression-Free Survival (PFS)
Description: Time to Progression-Free Survival (PFS) is the time from Baseline to the first Overall Response of Progressive Disease (PD) or death due to any cause if the subject dies without experiencing PD, calculated as date of first PD or date of death - date of Cycle 1 Day 1+1. PFS will be summarized in months, which will be obtained by dividing PFS in days by 30 days/month. Summary statistics will be determined using the KM estimate of the survival function for PFS. The between-treatment comparison will be performed using the logrank test.
Time Frame: From date of first treatment (Cycle 1 Day 1) until the date of first documented disease progression or date of death, which occurred first, assessed up to 36 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
months | 2.5 [1.8 to 6.1] | 1.9 [1.8 to 3.8]
Statistical Analysis 1: Comparison: CF102 vs Placebo Tablets of CF102; The between-treatment comparison (CF102 vs Placebo) will be performed on Time to Progression Free Survival using the logrank test; Test type: Other; p = 0.521, Log Rank

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is assessed as the percentage of subjects who achieved a Complete Response (CR) or Partial Response (PR). Per RECIST criteria v1.1, CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm; PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response is the sum of subjects achieving CR or PR.
Time Frame: The end of even-numbered cycles (Cycle 3 Day 1,Cycle 5 Day 1,Cycle 7 Day 1, Cycle 9 Day 1, Cycle 11 Day 1) assessed up to 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
Participants
  Cycle 3 Day 1 | 1 | 0
  Cycle 5 Day 1 | 2 | 0
  Cycle 7 Day 1 | 2 | 0
  Cycle 9 Day 1 | 2 | 0
  Cycle 11 Day 1 | 2 | 0

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is assessed as the percentage of subjects who achieved a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) using RECIST criteria. Per RECIST criteria v1.1, CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm; PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm) taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
Participants
  Cycle 3 Day 1 | 19 | 10
  Cycle 5 Day 1 | 9 | 2
  Cycle 7 Day 1 | 7 | 2
  Cycle 9 Day 1 | 5 | 2
  Cycle 11 Day 1 | 4 | 1

6. Secondary Outcome: Summary Statistics of Laboratory Parameters Associated With Viral Hepatitis, Hepatic Dysfunction, and Cirrhosis
Description: The raw and change from baseline (CFB) for each laboratory parameter (alanine aminotransferase (ALT), albumin, aspartate aminotransferase (AST), bilirubin (direct and total), International Normalized Ratio (INR),and prothrombin time (PT)) will be summarized by treatment and visit. CFB is calculated as (Value at Post-Baseline visit - Value at Baseline). The baseline value used in the calculations of CFB is the value taken at Cycle 1 Day 1.
Time Frame: Baseline (Cycle 1 Day 1); Cycle 11 Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 50 | 28
U/L
  ALT - Pre-Study: number analyzed (Participants) | 49 | 28
  ALT - Pre-Study | 47.4 (29.97) | 36.3 (20.93)
  ALT - Cycle 1 Day 1 | 46.5 (25.60) | 35.7 (26.75)
  ALT - Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  ALT - Cycle 11 Day 15 | 55.0 (45.39) | 44.0 (45.23)
  ALT - CFB to Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  ALT - CFB to Cycle 11 Day 15 | 7.2 (43.73) | 10.0 (23.17)
  AST - Pre-Study: number analyzed (Participants) | 49 | 28
  AST - Pre-Study | 83.8 (50.36) | 64.5 (38.49)
  AST - Cycle 1 Day 1 | 88.8 (58.88) | 66.7 (40.84)
  AST - Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  AST - Cycle 11 Day 15 | 77.1 (57.5) | 46.5 (23.90)
  AST - CFB to Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  AST - CFB to Cycle 11 Day 15 | 7.4 (46.34) | 8.3 (23.21)
  Albumin - Pre-Study: number analyzed (Participants) | 49 | 28
  Albumin - Pre-Study | 32.8 (4.97) | 33.7 (5.44)
  Albumin - Cycle 1 Day 1 | 32.4 (5.21) | 32.9 (5.50)
  Albumin - Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  Albumin - Cycle 11 Day 15 | 36.5 (3.88) | 35.8 (4.27)
  Albumin - CFB to Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  Albumin - CFB to Cycle 11 Day 15 | 2.2 (5.17) | -0.8 (8.85)
  Bilirubin (Direct) - Pre-Study: number analyzed (Participants) | 49 | 27
  Bilirubin (Direct) - Pre-Study | 9.0 (7.33) | 5.4 (3.32)
  Bilirubin (Direct) - Cycle 1 Day 1: number analyzed (Participants) | 50 | 27
  Bilirubin (Direct) - Cycle 1 Day 1 | 9.6 (9.00) | 5.3 (3.71)
  Bilirubin (Direct) - Cycle 11 Day 15: number analyzed (Participants) | 10 | 4
  Bilirubin (Direct) - Cycle 11 Day 15 | 4.2 (2.39) | 3.3 (0.96)
  Bilirubin (Direct) - CFB to Cycle 11 Day 15: number analyzed (Participants) | 10 | 4
  Bilirubin (Direct) - CFB to Cycle 11 Day 15 | -0.7 (3.16) | 1.3 (2.5)
  Bilirubin (Total) - Pre-Study: number analyzed (Participants) | 49 | 28
  Bilirubin (Total) - Pre-Study | 20.5 (12.9) | 14.9 (6.39)
  Bilirubin (Total) - Cycle 1 Day 1 | 21.1 (15.94) | 15.1 (9.62)
  Bilirubin (Total) - Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  Bilirubin (Total) - Cycle 11 Day 15 | 14.3 (4.10) | 9.8 (2.87)
  Bilirubin (Total) - CFB to Cycle 11 Day 15: number analyzed (Participants) | 11 | 4
  Bilirubin (Total) - CFB to Cycle 11 Day 15 | 0.7 (5.41) | 2.0 (3.56)
  Prothrombin Time (PT) - Pre-Study: number analyzed (Participants) | 46 | 28
  Prothrombin Time (PT) - Pre-Study | 12.39 (1.85) | 12.08 (1.097)
  PT - Cycle 1 Day 1 | 12.17 (1.37) | 12.30 (1.33)
  PT - Cycle 11 Day 15: number analyzed (Participants) | 9 | 4
  PT - Cycle 11 Day 15 | 11.82 (1.128) | 11.70 (0.942)
  PT - CFB to Cycle 11 Day 15: number analyzed (Participants) | 9 | 4
  PT - CFB to Cycle 11 Day 15 | 0.08 (0.657) | 0.53 (1.212)
  International Normalized Ratio (INR) - Pre-Study: number analyzed (Participants) | 46 | 28
  International Normalized Ratio (INR) - Pre-Study | 1.19 (0.176) | 1.15 (0.114)
  INR - Cycle 1 Day 1 | 1.17 (0.141) | 1.19 (0.138)
  INR - Cycle 11 Day 15: number analyzed (Participants) | 9 | 4
  INR - Cycle 11 Day 15 | 1.11 (0.105) | 1.13 (0.096)
  INR - CFB to Cycle 11 Day 15: number analyzed (Participants) | 9 | 4
  INR - CFB to Cycle 11 Day 15 | -0.01 (0.078) | 0.05 (0.129)
Statistical Analysis 1: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of ALT will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.988, ANCOVA
Statistical Analysis 2: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of AST will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.989, ANCOVA
Statistical Analysis 3: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of Albumin will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.717, ANCOVA
Statistical Analysis 4: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of Bilirubin (direct) will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.891, ANCOVA
Statistical Analysis 5: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of Bilirubin (Total) will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.275, ANCOVA
Statistical Analysis 6: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of PT will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.549, ANCOVA
Statistical Analysis 7: Comparison: CF102 vs Placebo Tablets of CF102; Between-treatment comparisons of INR will be performed at Cycle 11 Day 15 using ANCOVA with CFB as the dependent variable and the Baseline value of the variable as the covariate; Test type: Other; p = 0.479, ANCOVA

7. Secondary Outcome: Summary Statistics of White Blood Cell (WBC) Adenosine A3 Receptor (A3AR) Expression and Clinical Response - WBC Adenosine A3 Receptor (A3AR) Expression
Description: Summary statistics for WBC adenosine A3 receptor (A3AR) expression and CFB in WBC A3AR expression will be provided by treatment and visit. A3AR mRNA expression in WBC was determined from blood collected to a PAXgene RNA tubes (Qiagen, Venlo, The Netherlands), using the QuantiGene Plex 2.0® assay (Thermo Fisher, Waltham, MA, USA). β-actin was used as a reference control, and the oligonucleotide probe sets were designed by Thermo Fisher. Luminescence from each specific probe set was captured by Glomax Multi (Promega, Madison, WI, USA). A3AR was expressed in units, where 1 unit was defined as the mean of A3AR expression in healthy subjects (n = 50). Healthy subjects were 20-70 years of age with no known illness and no prior treatment.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 11 Day 1
Population: The analysis of the secondary outcome measure was performed using data from selected study sites on subjects in the Intent-To-Treat (ITT) Population, defined as all subjects who received at least one dose of study medication (i.e., Safety Population) with any post-Baseline assessment recorded. Exclusion of subjects from the ITT Population was determined prior to unblinding. The selection of study sites for participation in the A3AR blood sampling was determined according to the protocol.
Measure: Mean (Standard Deviation); unit: ratio of patient to healthy control
Arm/Group | CF102 | Placebo Tablets of CF102
Number analyzed (Participants) | 32 | 20
ratio of patient to healthy control
  Baseline - Cycle 1 Day 1 | 1.789 (2.2103) | 2.339 (3.2906)
  Cycle 11 Day 1: number analyzed (Participants) | 9 | 2
  Cycle 11 Day 1 | 2.821 (3.8114) | 1.1 (0.0849)
  CFB to Cycle 11 Day 1: number analyzed (Participants) | 9 | 2
  CFB to Cycle 11 Day 1 | 0.757 (0.7948) | -0.3 (0.5798)

8. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - CL/F (L/h)
Description: Describe the PK parameter CL/F (L/h) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: The PK analysis was conducted on advanced hepatocellular carcinoma patients with Child Pugh class B cirrhosis who received 25 mg BID for 29 days.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | CF102
Number analyzed (Participants) | 45
L/h | 12.42 (57.83)

9. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - Vc/F (L)
Description: Describe the PK parameter Vc/F (L) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | CF102
Number analyzed (Participants) | 45
L | 254.20 (54.56)

10. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - Vp/F (L)
Description: Describe the PK parameter Vp/F (L) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | CF102
Number analyzed (Participants) | 45
L | 49.99 (16.33)

11. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - Vss/F (L)
Description: Describe the PK parameter Vss/F (L) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | CF102
Number analyzed (Participants) | 45
L | 309.56 (44.31)

12. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - Elimination Half-life (Hours)
Description: Describe the PK parameter Elimination half-life (hours) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | CF102
Number analyzed (Participants) | 45
hours | 18.39 (29.93)

13. Secondary Outcome: Pharmacokinetics (PK) Parameters of CF102 - AUC_0-12, Steady State (ng*h/mL)
Description: Describe the PK parameter AUC_0-12, steady state (ng*h/mL) of namodenoson in subjects with Child-Pugh Class B cirrhosis who received twice daily administration of namodenoson for 29 days in Study CF102-201HCC at Day 1 and Day 29. In order to use a model-based Bayesian analysis in these subjects, a population PK (PPK) model of namodenoson had to be first created with the rich namodenoson concentration data available from two previously conducted studies (healthy volunteers in CF102-101 receiving single doses of 1 to 40 mg; and advanced hepatocellular carcinoma patients in CF102-102HCC receiving 1 to 25 mg BID of namodenoson for 29 days).
Time Frame: Cycle 1 Days 1, 8 and 15; Cycle 2 day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | CF102
Number analyzed (Participants) | 45
ng*h/mL | 2012.54 (57.83)

ADVERSE EVENTS:
Time Frame: AEs were recorded for each subject at the start of Cycle 1 Day 1 visit and followed to the 28-day Follow-Up Visit (28 days post End of Dosing) for up to 1 year/ Open-Label (OL) Follow-Up Visit (28 days post OL End of Dosing) for an average of 1 year. For observed toxicity thought to be at least possibly related to study drug was not resolved by the 28-day Follow-Up Visit/OL Follow-Up Visit, the subject was followed until the event resolved or stabilized, for an average of up to 24 months.
Description: Serious adverse event classification based on the FDA regulatory definition of a serious AE.
Arm/Group | CF102 | Placebo Tablets of CF102
All-Cause Mortality (participants affected / at risk) | 34/50 | 24/28
Serious Adverse Events (participants affected / at risk) | 37/50 | 20/28
Other Adverse Events (participants affected / at risk) | 46/50 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF102 (N=50) | Placebo Tablets of CF102 (N=28)
Subileus (Gastrointestinal disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 3 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Disease Progression (General disorders) | 13 | 5
Chest pain (General disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Hepatic enzyme increased/ (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Malignant neoplasm progression/ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF102 (N=50) | Placebo Tablets of CF102 (N=28)
Anaemia (Blood and lymphatic system disorders) | 8 | 5
Abdominal Pain (Gastrointestinal disorders) | 9 | 3
Ascites (Gastrointestinal disorders) | 10 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 9 | 6
Vomiting (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 7 | 6
Chest pain (General disorders) | 2 | 3
Disease Progression (General disorders) | 14 | 5
Fatigue (General disorders) | 9 | 3
Oedema peripheral (General disorders) | 10 | 5
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 3
Blood thyroid stimulating hormone increased (Investigations) | 1 | 3
Tri-iodothyronine free decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 4 | 4
Weight increased (Investigations) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 1
Hepatic encephalopathy (Nervous system disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02128958/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT02128958/SAP_001.pdf